CLINICAL TRIAL: NCT02070432
Title: An Open-label Study to Investigate the Tolerability, Pharmacokinetics and Anti-tumour Effect Following Photodynamic Therapy (PDT) With Single-ascending Doses of LUZ11 in Patients With Advanced Head and Neck Cancer
Brief Title: Photodynamic Therapy With LUZ11 in Advanced Head and Neck Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luzitin SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUZ11-CDU-001; 2013-003133-14 (EudraCT Number)
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: LUZ11; head and neck cancer; photodynamic therapy; Redaporfin
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LUZ11 PDT (Experimental): Study consists of two phases, in each participant:
  1. Dose-finding phase with sequential periods in which single-ascending doses of LUZ11 will be titrated up to a dose that shows to be effective following photoirradiation of small spots of tumor surface.
  2. Final PDT session with the previously identified individual effective dose.
  Interventions: Drug: LUZ11

INTERVENTIONS:
Drug: LUZ11 — LUZ11 i.v. administration followed by laser light irradiation

SUMMARY:
This study will investigate the tolerability, recommended dose and pharmacokinetics of LUZ11 following photodynamic therapy (PDT) of patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
LUZ11 is a new photosensitizer for use in photodynamic therapy (PDT) of solid tumors, such as head and neck cancer. PDT with LUZ11 involves the intravenous administration of LUZ11 followed by irradiation of the target tumor with laser light of an appropriate wavelength. The light causes the drug to react with oxygen, which forms reactive oxygen species (ROS) locally and induces tumor cells death and damages the blood vessels of the tumor thus preventing it from receiving nutrients.

The primary objective of this study is to assess the tolerability of LUZ11 following single ascending doses of LUZ11. The secondary objectives of this study are to explore the LUZ11 dose that has anti-tumor effect following photoactivation and to determine LUZ11 pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or non-pregnant, non-breast feeding women
* Karnofsky performance status of 60% or greater
* Histologically confirmed recurrent/refractory squamous cell carcinoma of the head and neck
* Clearly visible tumor on the oral cavity or cutaneous surface

Exclusion Criteria:

* Known hypersensitivity to any of the formulation ingredients
* Known hypersensitivity to porphyrins
* Porphyria or other diseases exacerbated by light
* Tumors known to be eroding into a major blood vessel in or adjacent to the irradiation site
* Planned skin phototherapy session(s) within the study timeframe
* Planned surgical procedure within the study timeframe
* Coexisting ophthalmic disease likely to require slit-lamp examination within the study timeframe
* Existing therapy with a photosensitizing agent
* Unstable angina and/or congestive heart failure requiring hospitalization within 6 months prior to screening
* Myocardial infarction within 6 months prior to screening
* Contraindication to MRI with gadolinium
* Unacceptable laboratory abnormalities
* Clinically relevant 12-lead ECG abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to 21 days following each dose-finding PDT session, and up to 13 weeks following final PDT session

SECONDARY OUTCOMES:
Depth of Tumor Necrosis Assessed by Diffusion-Weighted Magnetic Resonance Imaging (MRI) with Gadolinium as a Measure of Anti-Tumor Efficacy | Up to 21 days after each dose-finding PDT session, and up to 13 weeks after final PDT session

OTHER OUTCOMES:
LUZ11 Maximum Plasma Concentration (Cmax), Area Under the Concentration-Time Curve (AUC), Elimination Half-Life (T½), Volume of Distribution (Vd) and Clearance (CL) | Prior to dose, immediately after dose, and at 0.08, 0.5, 0.75, 1, 3, 6, 12, 24, 48 and 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Luis Almeida, MD, PhD, Study Director — Luzitin SA
Locations (2):
- Portugal (2):
  - Hospital CUF Porto, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE (IPO-Porto), Porto